CLINICAL TRIAL: NCT01995058
Title: A Randomized Phase 2 Study of Cabozantinib (XL184) in Combination With Abiraterone in Chemotherapy Naïve Subjects With Bone-Metastatic Castration-Resistant Prostate Cancer (CRPC)
Brief Title: Combo of Cabozantinib With Abiraterone in Chemotherapy-Naïve Subjects With Bone-Metastatic CRPC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decided to close the study prior to completion of enrollment. This was a business decision and not based on the safety results of the study.
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XL184-210
Record Dates: First submitted 2013-11-14; First posted 2013-11-26 (Estimated); Results first posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer; Castration Resistant Prostate Cancer; Prostatic Neoplasms
Keywords: CRPC; castration resistant prostate cancer; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cabozantinib; abiraterone; Abiraterone Acetate; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1: Cabozantinib 40 mg + abiraterone with prednisone (Experimental): Cabozantinib 40 mg, by mouth daily (po QD), + abiraterone with prednisone
  Interventions: Drug: cabozantinib; Drug: abiraterone; Drug: prednisone
- Arm 2: Cabozantinib 20 mg + abiraterone and prednisone (Experimental): Cabozantinib 20 mg, by mouth daily (po QD), + abiraterone with prednisone
  Interventions: Drug: cabozantinib; Drug: abiraterone; Drug: prednisone
- Arm 3: Cabozantinib 20 mg (every other day) + abiraterone and prednisone (Experimental): Cabozantinib 20 mg every other day with abiraterone and prednisone
  Interventions: Drug: cabozantinib; Drug: abiraterone; Drug: prednisone
- Arm 4: Abiraterone and prednisone only (Active Comparator): Abiraterone with prednisone
  Interventions: Drug: abiraterone; Drug: prednisone

INTERVENTIONS:
Drug: cabozantinib
  Other Names: XL184
  Arms: Arm 1: Cabozantinib 40 mg + abiraterone with prednisone; Arm 2: Cabozantinib 20 mg + abiraterone and prednisone; Arm 3: Cabozantinib 20 mg (every other day) + abiraterone and prednisone
Drug: abiraterone
  Other Names: Zytiga(R); abiraterone acetate
Drug: prednisone

SUMMARY:
This study was conducted in subjects in chemotherapy-naïve subjects with bone-metastatic castration-resistant prostate cancer (CRPC).

DETAILED DESCRIPTION:
The goal of this clinical trial was to learn if the combination of the drugs cabozantinib and abiraterone works for men that were chemotherapy-naive, bone metastasis CRPC patients. It was designed to learn about the safety of cabozantinib. The main questions are:

1. Does it work and is it safe in men with chemotherapy-naïve bone- metastatic castration resistant CRPC?
2. What was the clinical benefit at different dose levels of the combination of abiraterone and cabozantinib in this patient population?

Participants were assigned to one of the four treatment groups:

Arm 1. cabozantinib at a dose of 40 mg every day (QD) plus abiraterone with prednisone; Arm 2. cabozantinib at a dose of 20 mg QD plus abiraterone with prednisone; Arm 3. cabozantinib at a dose of 20 mg every other day (QOD) plus abiraterone with prednisone; Arm 4. abiraterone with prednisone.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate.
* Must be surgically or medically castrated (serum testosterone levels less than or equal to 50 ng/dL)
* Must have castration-resistant prostate cancer (CRPC) with disease progression during LHRH therapy or after a surgical bilateral orchiectomy.
* Bone metastasis related to prostate cancer
* Adequate organ and marrow function
* Capable of understanding and complying with the protocol requirements and signed the informed consent document
* Sexually active subjects and their partners must agree to use medically accepted methods of barrier contraception (eg, male condom or female condom) as well as one other medically accepted method of contraception during the course of the study treatment and for 4 months after the last dose of study treatment.

Exclusion Criteria:

* Any prior treatment with abiraterone, enzalutamide, or any investigational agents blocking androgen receptor (AR) or androgen synthesis.
* Any prior treatment with cabozantinib or participation in a prior clinical trial of cabozantinib.
* Any prior cytotoxic therapy (including estramustine) or biologic therapy for the treatment of prostate cancer (a few exceptions will be allowed)
* Any prior radionuclide therapy (eg, samarium 153, strontium 89, alpharadin)
* Use of investigational agent within 28 days
* Any pathological finding consistent with small cell carcinoma of the prostate
* Known brain metastases or cranial epidural disease
* Diagnosis of another malignancy within 2 years, except for superficial non-melanoma skin cancers, or localized, low grade tumors deemed cured and not treated with systemic therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Scottsdale, Arizona
  - Sedona, Arizona
  - Tucson, Arizona
  - Oxnard, California
  - San Diego, California
  - Aurora, Colorado
  - Athens, Georgia
  - Atlanta, Georgia
  - Peoria, Illinois
  - Wichita, Kansas
  - Las Vegas, Nevada
  - Raleigh, North Carolina
  - Tualatin, Oregon
  - Charleston, South Carolina
  - Greenville, South Carolina
  - Myrtle Beach, South Carolina
  - Dallas, Texas
  - Houston, Texas
  - Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled subjects from 11 February 2014 (first patient enrolled) through 02 September 2014 (Sponsor decision to end study). The study was terminated prior to completing enrollment due to Sponsor decision (not based on any safety results).
Groups:
- Arm 1 - Cabozantinib 40 mg, po QD + Abiraterone: Cabozantinib 40 mg, po QD + abiraterone with prednisone
- Arm 2 - Cabozantinib 20 mg, po QD + Abiraterone: Cabozantinib 20 mg, po QD + abiraterone with prednisone
- Arm 3 - Cabozantinib 20 mg, po QOD + Abiraterone: Cabozantinib 20 mg, po QOD + abiraterone with prednisone
- Arm 4 - Abiraterone Only: Abiraterone with prednisone
Period: Overall Study
Arm/Group | Arm 1 - Cabozantinib 40 mg, po QD + Abiraterone | Arm 2 - Cabozantinib 20 mg, po QD + Abiraterone | Arm 3 - Cabozantinib 20 mg, po QOD + Abiraterone | Arm 4 - Abiraterone Only
Started (Randomized) | 14 | 13 | 13 | 14
Completed (Subjects still on study treatment as of the data cut-off date) | 0 | 0 | 0 | 0
Not Completed | 14 | 13 | 13 | 14
Not completed — Sponsor Decision to terminate study | 14 | 12 | 12 | 10
Not completed — Progressive Disease | 0 | 1 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1
Not completed — No Treatment Given | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm 4 - Abiraterone Only: Abiraterone with prednisone only
- Total: Total of all reporting groups
Arm/Group | Arm 1 - Cabozantinib 40 mg, po QD + Abiraterone | Arm 2 - Cabozantinib 20 mg, po QD + Abiraterone | Arm 3 - Cabozantinib 20 mg, po QOD + Abiraterone | Arm 4 - Abiraterone Only | Total
Number analyzed (Participants) | 14 | 13 | 13 | 14 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 3 | 3 | 10
  >=65 years | 12 | 11 | 10 | 11 | 44
Age, Continuous [Median (Full Range); unit: years] | 76 [56 to 87] | 74 [61 to 83] | 73 [63 to 76] | 70 [55 to 84] | 73 [55 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 14 | 13 | 13 | 14 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 12 | 13 | 14 | 52
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 3 | 2 | 8
  White | 13 | 10 | 10 | 12 | 45
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 13 | 13 | 14 | 54

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Progression Free Survival (PFS)
Description: PFS is defined as the time from randomization to the earlier of disease progression or death due to any cause, as assessed by Independent Radiology Committee (IRC). The sponsor terminated the study early due to business reasons. As such, no data were collected for efficacy analyses.
Time Frame: Up to 18 Months
Population: As pre-specified in the protocol, a total of 140 PFS events were required for this analysis; given that only 54 participants were enrolled and the study terminated early after 9 months, no data were collected or analyzed as planned for this outcome measure.
Arm/Group | Arm 1 - Cabozantinib 40 mg, po QD + Abiraterone | Arm 2 - Cabozantinib 20 mg, po QD + Abiraterone | Arm 3 - Cabozantinib 20 mg, po QOD + Abiraterone | Arm 4 - Abiraterone Only
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 7 months
Description: One subject was randomized to the 20 mg QOD combination arm but received 20 mg cabozantinib treatment on a QD schedule according to the clinical database dosing records. In the Safety population, this subject was included in the 20 QD combination arm and not in the 20 QOD combination arm. Another subject was randomized to the abiraterone only arm, but never received study treatment.
Groups:
- Arm 1: Cabozantinib 40 mg, po QD + abiraterone with prednisone
- Arm 2: Cabozantinib 20 mg, po QD + abiraterone with prednisone
- Arm 3: Cabozantinib 20 mg, po QOD + abiraterone with prednisone
- Arm 4: Abiraterone with prednisone
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
All-Cause Mortality (participants affected / at risk) | 0/14 | 1/14 | 0/12 | 1/13
Serious Adverse Events (participants affected / at risk) | 2/14 | 4/14 | 1/12 | 1/13
Other Adverse Events (participants affected / at risk) | 13/14 | 10/14 | 11/12 | 11/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=14) | Arm 2 (N=14) | Arm 3 (N=12) | Arm 4 (N=13)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uncoded: left sided obstructive uropathy (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Mucositis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural hematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uncoded: swelling to left tongue (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=14) | Arm 2 (N=14) | Arm 3 (N=12) | Arm 4 (N=13)
Hypertension (Vascular disorders) | 3 (3) | 3 (3) | 3 (3) | 2 (2)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lip pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 4 (4) | 3 (3) | 2 (2) | 3 (3)
Feeling abnormal (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical device complication (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
White blood cell count decreased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 2 (2) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 4 (4)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Mood altered (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 1 (1) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pallor (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Systolic hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uncoded: BILATERAL ANKLE EDEMA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uncoded: HYPOTENSION AND DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uncoded: PAIN IN CHEST/NECK/LOWER JAW (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uncoded: PAIN - LEFT SHOULDER, SCAPULA, NECK (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uncoded: PAIN-BILATERAL RIBS, KNEES, LEFT ANKLE (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uncoded: R. FOOT SLAPPING DOWN WHEN WALKING (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated for business reasons prior to completing enrollment. No efficacy data were collected and limited safety data were collected. No statistical comparisons between treatment arms could be made due to low subject numbers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreements with investigators vary; constant is our right to review results communications prior to public release, and embargo communications for a period of ≤60 days from submittal for review. We do not prohibit investigators from publishing, but we may require previously undisclosed confidential information, other than study results, to be removed from publications, and single-center publications are postponed until after publication of the trial's primary multicenter publication.